CLINICAL TRIAL: NCT06470971
Title: Immune Checkpoint Inhibitor Rechallenge in Combination With Siltuximab Prophylaxis for Patients Who Had Prior Immune-Related Adverse Event (CIRES Trial)
Brief Title: Siltuximab for the Prevention of Severe Immune-Related Adverse Events During Immune Checkpoint Inhibitor Rechallenge in Patients With Advanced Cancer, CIRES Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yuanquan Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanquan Yang, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-23393; NCI-2024-04853 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — spartalizumab; Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PD1 antibody, PD-L1 antibody, Siltuximab) (Experimental): Patients receive anti-PD1 or anti-PD-L1 monoclonal antibody therapy either every 3 or 6 weeks, or every 2 or 4 weeks per physicians choice. Patients also receive siltuximab IV over 1 hour on day 1 of each cycle prior to the administration of anti-PD1 or anti-PD-L1 therapy. Treatment repeats either every 3 weeks for up to 8 doses or every 4 weeks for up to 6 doses in the absence of disease progression or unacceptable toxicity. Patients may undergo biopsy and bone scan on study, as well as blood sample collection and CT or MRI throughout the study.
  Interventions: Biological: Anti-PD-L1 Monoclonal Antibody; Biological: Anti-PD1 Monoclonal Antibody; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Biological: Siltuximab

INTERVENTIONS:
Biological: Anti-PD-L1 Monoclonal Antibody — Receive anti-PD-L1 monoclonal antibody therapy
Biological: Anti-PD1 Monoclonal Antibody — Receive anti-PD1 monoclonal antibody therapy
  Other Names: Anti-PD-1 Monoclonal Antibody
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Siltuximab — Given IV
  Other Names: Anti-IL-6 Chimeric Monoclonal Antibody; cCLB8; CNTO 328; CNTO-328; Sylvant

SUMMARY:
This phase II trial studies how well giving siltuximab during the reintroduction (rechallenge) of immune checkpoint inhibitor (ICI) therapy works in preventing severe immune-related adverse events (irAEs) in patients with cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Immune checkpoint inhibitors, such as anti-PD1 and anti-PD-L1 monoclonal antibodies, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The use of ICI therapy may lead to severe irAEs that can affect essentially any organ system in the body. Severe irAEs may lead to the early stopping of life saving treatment. Most patients that stop ICI therapy early will eventually progress and require additional treatment. Sometimes the decision is made to rechallenge with ICI therapy. Many patients who developed severe irAEs during initial ICI therapy are at risk for developing severe irAEs again during the rechallenge. Siltuximab is a monoclonal antibody that binds to receptors for a protein called interleukin-6 (IL-6). This may help lower the body's immune response and reduce inflammation. Giving siltuximab during ICI rechallenge may help prevent severe irAEs in patients with advanced cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether siltuximab prophylaxis reduces rates of de novo or recurrent severe irAE within 24 weeks of anti-PD-1/PD-L1 therapy rechallenge.

SECONDARY OBJECTIVE:

I. To assess the preliminary anti-tumor activity of this combination including overall response rate (ORR), progression-free survival (PFS) and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To evaluate potential predictive biomarkers such as baseline serum IL-6 level, C-reactive protein (CRP) suppression level, tissue IL-6 expression, stool microbiome, and antibody clearance rate.

II. To assess changes in immune cell infiltration of irAE site pre- and post-treatment by multiomics profiling.

III. To assess patient-reported outcomes by Patient-Reported Outcomes Measurement Information System (PROMIS) instruments.

IV. To correlate circulating tumor deoxyribonucleic acid (ctDNA) levels with treatment responses.

OUTLINE:

Patients receive anti-PD1 or anti-PD-L1 monoclonal antibody therapy either every 3 or 6 weeks, or every 2 or 4 weeks per physicians choice. Patients also receive siltuximab intravenously (IV) over 1 hour on day 1 of each cycle prior to the administration of anti-PD1 or anti-PD-L1 therapy. Treatment repeats either every 3 weeks for up to 8 doses or every 4 weeks for up to 6 doses in the absence of disease progression or unacceptable toxicity. Patients may undergo biopsy and bone scan on study, as well as blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at day 28, every 12 weeks for up to 2 years, and then every 6 months until 5 years following registration.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients with any advanced cancer types who would benefit from anti-PD1 or anti-PD-L1 therapy rechallenge at the investigator's discretion
* Patients must have had prior severe irAE while on ICI monotherapy or in combination with other anticancer treatment. Severe irAE is defined as any grade 2 or higher irAE requiring treatment discontinuation and prednisone > 0.5 milligrams (mg)/kilogram (kg)/day (or equivalent) followed by a taper ≥ 4 weeks. Patients with history of grade 4 severe irAE need to carefully weigh the risks and benefits and might be eligible on a case-by-case basis after discussion with principal investigator (PI)
* Recovery from prior irAEs to ≤ grade 1
* Patients who are on prednisone ≤ 10 mg/day (d) or equivalent are allowed
* Hemoglobin > 7 g/dL and < 17 g/dL
* Absolute neutrophil count (ANC) ≥ 1000 per mm^3
* Platelet count ≥ 75 × 10^9/L
* Serum bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN or ≤ 5 × ULN for patients with liver metastases
* Measured or calculated creatinine clearance (CL) ≥ 30 mL/min except patients with end-stage renal disease on hemodialysis
* Cycle 1 day 1 of the study treatment should be at least 2 weeks since prior systemic therapy, radiotherapy, or surgery
* Estimated life expectancy, in the judgment of the investigator, of at least 12 weeks
* Subjects of childbearing potential must have a negative serum pregnancy test at screening
* Subjects of childbearing potential must be willing to completely abstain or agree to use a highly effective method of contraception (i.e., less than 1% failure rate), from the time of signing informed consent and for the duration of study participation through 3 months following the last dose of study drug

  * Childbearing potential is defined by the following criteria: 1. Subject has not undergone a hysterectomy or bilateral oophorectomy; or 2. has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
  * Highly effective birth control methods (less than 1% failure rate per year if used consistently and correctly) include but are not limited to: 1. Oral, injected, or implanted hormonal method of contraception; 2. Place of intrauterine device (IUD) or system (IUS); 3. Tubal ligation (tubes tied) or a sterile partner (effective bilateral vasectomy)
* Subjects must not breastfeed a child during the study and for 3 months after the last dose of study drug
* Ability to understand and willingness to sign the written informed consent document

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Any ≥ grade 3 irAEs in which the risks outweigh the benefits per investigator's discretion (these may include but are not limited to myocarditis, myasthenia gravis, Guillain-Barré syndrome, encephalitis, myelitis, or other life-threatening events)
* Has active autoimmune disease or irAE requiring systemic treatment with steroids (> 10 mg daily doses of prednisone or equivalent) or other immunosuppressive agents or any condition that, in the investigator's judgment, precludes treatment with anti-PD-1/PD-L1 therapy
* Cycle 1 day 1 of the study treatment must be at least 2 weeks beyond high dose systemic corticosteroids (prednisone > 0.5 mg/kg/day or equivalent); chronic steroid use up to 10 mg daily prednisone (or equivalent) is permitted
* Other concurrent anticancer therapy except for palliative radiation and hormone therapy
* Has a known history of HIV-1/2 with detectable viral load and/or CD4 (cluster of differentiation 4) count < 300/mL within the previous 3 months
* Has detectable hepatitis B virus (HBV) or hepatitis C virus (HCV) viral load polymerase chain reaction (PCR) if there is a known history of active hepatitis B or hepatitis C
* High risk for bowel perforation per the investigator's judgment, such as history of severe diverticulitis or active ulcers or extensive gastrointestinal (GI) involvement by the tumor
* Presence of a transplanted solid organ (with the exception of a corneal transplant more than 3 months prior to screening) or having received an allogeneic bone marrow transplant or an allogeneic peripheral blood stem cell transplant
* Uncontrolled concomitant illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, myocardial infarction within 1 month prior to enrollment, uncontrolled cardiac arrhythmias, uncontrolled seizures, or severe noncompensated hypertension (systolic blood pressure > 180mmHg or diastolic blood pressure > 120mmHg)
* Patients with a current severe infection
* Known unmanageable allergies, hypersensitivity, intolerance to monoclonal antibodies, to murine, chimeric, human proteins or their excipients
* Prior failure of interleukin-6 or interleukin-6 receptor targeted therapies. Prior IL-6 or IL-6 receptor-targeted therapies are permitted if the response was favorable
* Received any investigational drug within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe immune-related adverse event (irAE) | Within 24 weeks of immune checkpoint inhibitor (ICI) rechallenge
  Will be assessed per National Cancer Institute Common Terminology Criteria for Adverse Events version (v) 5.0. irAEs are defined as AEs of immune nature (i.e., inflammatory) in the absence of a clear alternative etiology. The investigators will determine if an AE should be classified as irAE (yes/no). Will be defined as ≥ grade 2 requiring treatment discontinuation and prednisone > 0.5 milligrams/kilogram/day or equivalent followed by a taper ≥ 4 weeks) within 24 weeks of ICI rechallenge.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years
  Will be determined per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Will be calculated as the percentage of patients achieving complete response or partial response. The exact binomial 95% confidence interval (CI) will be provided.
Median progression-free survival | Initiation of therapy to time of progression or death, whichever occurs first, assessed up to 5 years
  Will be determined per RECIST v1.1. Survival will be analyzed using Kaplan-Meier methods, resulting in median survival times with 95% CI.
Overall survival | Initiation of therapy to death, assessed up to 5 years
  Will be determined per RECIST v1.1. Survival will be analyzed using Kaplan-Meier methods, resulting in median survival times with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanquan Yang, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu